CLINICAL TRIAL: NCT04487678
Title: A Single-centre, Randomised, Single-blinded Crossover Study Evaluating the Metabolic Effects of a Ketone Ester Food Supplement in People With Type 1 Diabetes
Brief Title: Exogenous Ketones in People With Type 1 Diabetes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Prioritization of other projects
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: KEsupplements
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Ketosis, Diabetic
MeSH Terms: conditions — Diabetic Ketoacidosis

STUDY DESIGN:
Intervention Model Description: Single-centre, randomised, single blinded, crossover study in 6 individuals with type 1 diabetes (see inclusion/exclusion criteria)
Who Masked: Participant
Masking Description: There will be two intervention arms that will take place in a randomised, single blinded fashion so that participants are not aware of which dose of ketone esters they receive
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-dose KE (Experimental): 141 mg/kg bodyweight of ketone esters
  Interventions: Dietary Supplement: Ketone ester supplement
- High-dose KE (Experimental): 282 mg/kg bodyweight of ketone esters
  Interventions: Dietary Supplement: Ketone ester supplement

INTERVENTIONS:
Dietary Supplement: Ketone ester supplement — Participants taking part in this study will receive a drink containing either 141 or 282 mg/kg bodyweight of ketone esters in a randomised order. These doses are in line with recommendations by the company HVMN from which the supplements for this study will be obtained.
  Other Names: H.V.M.N Ketone Ester food supplement

SUMMARY:
The aim of this pilot study is to investigate the metabolic effects of exogenous ketone ester food supplements, by assessing the change in blood acid-base balance, and the level of blood beta-hydroxy-butyrate in people with type 1 diabetes during resting conditions.

DETAILED DESCRIPTION:
The ketone bodies acetoacetate, β-hydroxybutyrate (βHB) and acetone are small lipid-derived molecules that are produced in the liver under certain conditions such as starvation, very low carbohydrate intake and prolonged glycogen-depleting exercise. Ketone bodies serve as an alternative energy substrate for the brain and other metabolically active tissues under periods of low glucose availability, and can modulate carbohydrate and lipid metabolism. Previously, controlled physiological ketosis required a low carbohydrate diet, starvation or administration of acetoacetate (AcAc) salts which were all unpleasant or potentially harmful. The development of ketone esters provides an alternative method to increase βHB levels, and has been shown to be well tolerated in rodents and humans. Two examples are the R,S-1,3-butanediol acetoacetate diester and the (R)-3-hydroxybutyl (R)-3-hydroxybutyrate ketone monoester. Ingestion of either have been shown to result in short-term (0.5-6 hours) nutritional ketosis (βHB >1mM). Nutritional ketosis can therefore be achieved without the need for the impracticality of ketogenic dieting or fasting.

In recent years there has been considerable interest in ketone body food supplements due to their potential for improved exercise performance and therapeutic glucose lowering effects in people with type 2 diabetes. Exogenous ketone supplements may be of particular interest for individuals living with type 1 diabetes by serving as an alternative fuel substrate to reduce the reliance on glucose utilisation and spare endogenous glycogen and reduce the risk of hypoglycaemia in certain situations, such as exercise. Stubbs et al. (2017) found that drinks containing exogenous ketones were a practical and efficacious way to raise blood βHB levels with only a modest change in acid-base balance in healthy individuals without diabetes (after 60 min, blood pH declined from 7.41 to 7.31 following a ketone ester drink). To date, no studies have investigated the metabolic effects of ketone in people with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for >1 year
* Male and female aged 18-45 years old
* HbA1c <8.5% (69 mmol/mol) based on analysis from the central laboratory unit of Bern University Hospital
* Using either continuous subcutaneous insulin infusion or multiple daily injections
* Wearing a continuous glucose monitor (CGM) or flash glucose monitor (fGM)
* Written informed consent

Exclusion Criteria:

* Physical or psychological disease likely to interfere with the normal conduct of the study and interpretation of the results as judged by the investigator
* Current treatment with drugs known to interfere with metabolism e.g. systemic corticosteroids, statins, SGLT2 inhibitors, GLP1 agonists
* Relevant diabetic complications as judged by the investigator
* Body mass index > 30 kg/m2
* Uncontrolled hypertension (>180/100 mmHg)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Males
Enrollment: 0 (Actual)
Dates: Start 2023-08 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in venous blood pH | Over a 3 hour period from baseline following ingestion of a ketone ester drink in people with type 1 diabetes.
  Change in blood pH over a 3 hour period from baseline following ingestion of a ketone ester drink

SECONDARY OUTCOMES:
Blood total ketone level /beta hydroxy butyrate level | 3 hours
Blood glucose concentration | 3 hours
Substrate oxidation rates determined using indirect calorimetry, via RER (respiratory exchange ratio) | 3 hours
Gastro-intestinal distress symptoms via a questionnaire | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Stettler, MD, Principal Investigator — University of Bern

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balasse EO, Fery F. Ketone body production and disposal: effects of fasting, diabetes, and exercise. Diabetes Metab Rev. 1989 May;5(3):247-70. doi: 10.1002/dmr.5610050304. PMID 2656155
- [Background] Clarke K, Tchabanenko K, Pawlosky R, Carter E, Todd King M, Musa-Veloso K, Ho M, Roberts A, Robertson J, Vanitallie TB, Veech RL. Kinetics, safety and tolerability of (R)-3-hydroxybutyl (R)-3-hydroxybutyrate in healthy adult subjects. Regul Toxicol Pharmacol. 2012 Aug;63(3):401-8. doi: 10.1016/j.yrtph.2012.04.008. Epub 2012 May 3. PMID 22561291
- [Background] Cox PJ, Clarke K. Acute nutritional ketosis: implications for exercise performance and metabolism. Extrem Physiol Med. 2014 Oct 29;3:17. doi: 10.1186/2046-7648-3-17. eCollection 2014. PMID 25379174
- [Background] Cox PJ, Kirk T, Ashmore T, Willerton K, Evans R, Smith A, Murray AJ, Stubbs B, West J, McLure SW, King MT, Dodd MS, Holloway C, Neubauer S, Drawer S, Veech RL, Griffin JL, Clarke K. Nutritional Ketosis Alters Fuel Preference and Thereby Endurance Performance in Athletes. Cell Metab. 2016 Aug 9;24(2):256-68. doi: 10.1016/j.cmet.2016.07.010. Epub 2016 Jul 27. PMID 27475046
- [Background] Egan B. The glucose-lowering effects of exogenous ketones: is there therapeutic potential? J Physiol. 2018 Apr 15;596(8):1317-1318. doi: 10.1113/JP275938. Epub 2018 Mar 24. No abstract available. PMID 29473164
- [Background] Egan B, D'Agostino DP. Fueling Performance: Ketones Enter the Mix. Cell Metab. 2016 Sep 13;24(3):373-375. doi: 10.1016/j.cmet.2016.08.021. PMID 27626197
- [Background] Evans M, Cogan KE, Egan B. Metabolism of ketone bodies during exercise and training: physiological basis for exogenous supplementation. J Physiol. 2017 May 1;595(9):2857-2871. doi: 10.1113/JP273185. Epub 2016 Dec 7. PMID 27861911
- [Background] Flint A, Raben A, Blundell JE, Astrup A. Reproducibility, power and validity of visual analogue scales in assessment of appetite sensations in single test meal studies. Int J Obes Relat Metab Disord. 2000 Jan;24(1):38-48. doi: 10.1038/sj.ijo.0801083. PMID 10702749
- [Background] Kesl SL, Poff AM, Ward NP, Fiorelli TN, Ari C, Van Putten AJ, Sherwood JW, Arnold P, D'Agostino DP. Effects of exogenous ketone supplementation on blood ketone, glucose, triglyceride, and lipoprotein levels in Sprague-Dawley rats. Nutr Metab (Lond). 2016 Feb 4;13:9. doi: 10.1186/s12986-016-0069-y. eCollection 2016. PMID 26855664
- [Background] Myette-Cote E, Neudorf H, Rafiei H, Clarke K, Little JP. Prior ingestion of exogenous ketone monoester attenuates the glycaemic response to an oral glucose tolerance test in healthy young individuals. J Physiol. 2018 Apr 15;596(8):1385-1395. doi: 10.1113/JP275709. Epub 2018 Mar 2. PMID 29446830
- [Background] Pinckaers PJ, Churchward-Venne TA, Bailey D, van Loon LJ. Ketone Bodies and Exercise Performance: The Next Magic Bullet or Merely Hype? Sports Med. 2017 Mar;47(3):383-391. doi: 10.1007/s40279-016-0577-y. PMID 27430501
- [Background] Robinson AM, Williamson DH. Physiological roles of ketone bodies as substrates and signals in mammalian tissues. Physiol Rev. 1980 Jan;60(1):143-87. doi: 10.1152/physrev.1980.60.1.143. No abstract available. PMID 6986618
- [Background] Stubbs BJ, Cox PJ, Evans RD, Santer P, Miller JJ, Faull OK, Magor-Elliott S, Hiyama S, Stirling M, Clarke K. On the Metabolism of Exogenous Ketones in Humans. Front Physiol. 2017 Oct 30;8:848. doi: 10.3389/fphys.2017.00848. eCollection 2017. PMID 29163194